CLINICAL TRIAL: NCT03599193
Title: A Randomized, Open-Label, Multiple Dose, Bioavailability Study of DFD-03 (Tazarotene Lotion, 0.1 % ) Dosed Twice Daily Compared to Once Daily Tazorac® (Tazarotene) Cream, 0.1% in Patients With Moderate Acne Vulgaris
Brief Title: A Bioavailability Study of DFD-03 Compared to Tazorac® in Patients With Moderate Acne Vulgaris
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DFD-03-CD-007
Record Dates: First submitted 2018-06-29; First posted 2018-07-26 (Actual); Results first posted 2020-09-14 (Actual); Last update posted 2021-03-01 (Actual); Status verified 2021-02

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Tazarotene and tazarotenic acid plasma concentrations will be determined at a designated laboratory from the blinded samples using a validated bioanalytical method.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- DFD-03 Lotion (Experimental): DFD-03 Lotion will be applied to the affected areas twice daily for 1 minute and rinsed off. 29 subjects will be enrolled into this arm.
  Interventions: Drug: Tazarotene Lotion, 0.1%
- Tazorac Cream (Active Comparator): Tazorac Cream will be applied to the affected areas once daily and left on for ~12 hours. 29 subjects will be enrolled into this arm.
  Interventions: Drug: Tazarotene Cream, 0.1%

INTERVENTIONS:
Drug: Tazarotene Lotion, 0.1% — DFD-03 (Tazarotene Lotion, 0.1%) applied Twice Daily for 1 minute and rinsed off
  Other Names: DFD-03 Lotion
  Arms: DFD-03 Lotion
Drug: Tazarotene Cream, 0.1% — Tazorac® (tazarotene) Cream, 0.1% applied Once Daily and left for approximately 12 hours
  Other Names: Tazorac Cream
  Arms: Tazorac Cream

SUMMARY:
This was a multicenter, randomized, multiple-dose, laboratory-blinded, open-label, 2-arm, parallel-arm study in subjects with moderate acne vulgaris.

DETAILED DESCRIPTION:
This was a multicenter, randomized, multiple-dose, laboratory-blinded, open-label, 2-arm, parallel-arm study in subjects with moderate acne vulgaris.

Approximately 62 subjects were randomized, stratified by age (Adult subjects: 17 years or older; Pediatric subjects: 9 years to 16 years 11 months for the Test product and 12 years to 16 years 11 months for the Reference product). The study was conducted in two parts, Part A and Part B in a sequential manner. Based on full PK profiles generated for adult subjects in Part A, the sparse PK sampling design in pediatric population was established in Part B.

ELIGIBILITY:
Inclusion Criteria:

1. Subject understands the study procedures, is willing to comply with the study procedures and required visits, and agrees to participate by giving written informed consent. Subjects under the legal age of consent must provide written assent and must have the written informed consent of their legal guardian.
2. Subject (or legal guardian) must be willing to authorize use and disclosure of protected health information collected for the study.
3. Male or female at least 9 years of age for the DFD-03 (Test) group and at least 12 years of age for the Tazorac Cream (Reference) group.
4. Female subjects must be having their menstrual period at Baseline (Day 1, as reported by the subject), except for subjects using hormonal contraceptives that preclude menstrual periods, if the subject is premenarcheal, is postmenopausal for at least 12 months prior to baseline, is surgically sterilized (i.e., tubal ligation) or if the subject is without a uterus and/or both ovaries.
5. A clinical diagnosis of facial acne vulgaris with a facial Investigator's Global Assessment (IGA) score of 3 (moderate) at Baseline (Day 1).
6. Subjects should have acne lesions on at least 1 of the following regions at the Screening visit: neck, upper chest, upper back (including shoulders).

   • This criterion is not applicable to the 9-11 years and 11 months age group.
7. Inflammatory lesion count (papules and pustules) of at least 20 on the face, including the nose, at Baseline (Day 1).

   • This criterion is not applicable to the 9-11 years and 11 months age group.
8. Non-inflammatory lesion count (closed and open comedones) of at least 25 on the face, including the nose, at Baseline (Day 1).

   • This criterion is not applicable to the 9-11 years and 11 months age group.
9. No more than 2 nodulocystic lesions on the face, including the nose, at Baseline (Day 1).
10. Females, regardless of childbearing potential:

    1. Must have a negative serum pregnancy test at Screening and a negative urine pregnancy test at Baseline (Day 1). Urine pregnancy test must have a sensitivity of at least 25 mIU/mL for βhCG.
    2. If sexually active, must be on or use an acceptable method of birth control. Acceptable methods of birth control include hormonal methods* or intrauterine device in use ≥ 90 days prior to Baseline (Day 1); or partner has had a vasectomy at least 90 days prior to Baseline (Day 1); or barrier methods plus spermicide; or Essure® that has been in place for at least 3 months before the screening visit with radiograph confirmation of fallopian tube blockage.

       * Hormonal methods: If on hormonal contraceptives, must have been on the same hormonal contraceptive product for 3 months (90 days) prior to Baseline (Day 1) and continued on same method and dose throughout the duration of the study. If subject had used hormonal birth control and had stopped, this should have occurred more than 6 months prior to Baseline.

    Exception: Sexually inactive female subjects are not required to practice a reliable method of contraception and may be enrolled at the investigator's discretion if they are counseled to remain sexually inactive for the duration of the study and understand the possible risks involved in getting pregnant during the study. An abstinent female must agree that if she becomes sexually active during the study she will use an acceptable form of contraception such as a barrier method with spermicide.
11. Subjects agree not to use any product on the face during the entire course of study except for non-medicated, investigator-approved cleanser, sunscreen, face wash, and make-up. Subjects should continue to use these investigator-approved products for the duration of the study and should avoid any changes in these consumer products.
12. Subjects must be willing to comply with sun avoidance measures for the face (as well as back/chest and shoulders, if applicable) including use of investigator-approved sunscreen and/or hats, have limited direct sunlight exposure time, and have no tanning bed use or use of other UV light sources during participation in the study.
13. Subject must be in good general health as determined by the investigator and supported by the medical history, physical examination, and normal or not clinically significant abnormal vital signs (blood pressure and pulse).

Exclusion Criteria:

1. Females who are pregnant or lactating or planning to become pregnant during the study period.
2. Treatment with the following products:

   1. Topical acne treatments (other retinoids, antibiotics, benzoyl peroxide, azelaic acid, resorcinol, salicylates, α-hydroxy/glycolic acid), or other topical facial medication (antifungals, steroids, anti-inflammatories) on the treatment area in the 14 days prior to Baseline (Day 1), including prescription and non-prescription products.
   2. Systemic corticosteroids, systemic acne treatments including systemic antibiotics used for treatment of acne, potential photosensitizing agents (thiazides, phenothiazines), spironolactone, flutamide, or immunosuppressant drugs in the 30 days prior to Baseline (Day 1).
   3. Systemic retinoid use (including high-dose vitamin A > 10,000 units per day) in the 180 days prior to Baseline (Day 1).
   4. Undertaken certain facial procedures such as chemical peel, laser treatment, photodynamic therapy, acne surgery, cryodestruction or chemodestruction, x-ray therapy, intralesional steroids, dermabrasion, or depilation (except eyebrow shaping) in the 30 days prior to Baseline (Day 1). After the subject is enrolled in the study, eyebrow shaping (except for tweezing) is prohibited.
   5. Treatment with a medication or procedure that, in the opinion of the investigator, would put the subject at unacceptable risk for participation in the study or may interfere with evaluations in the study.
   6. Treatment with an investigational product or device in the 30 days prior to Baseline (Day 1).
3. Known allergic reaction to retinoids or tazarotene or any of the other ingredients of these products. The inactive ingredients are sodium lauryl sulphate, stearyl alcohol, cetyl alcohol, gluconolactone, Vitamin E polyethylene glycol succinate, glycerin, carbomer P 971, propylparaben, methylparaben, edetate disodium, butylated hydroxytoluene, medium-chain triglyceride, trolamine, and purified water.
4. Presence of any facial skin disease or condition that would interfere with the study or place the subject at unacceptable risk including sunburn, rosacea, seborrheic dermatitis, perioral dermatitis, lupus, dermatomyositis, psoriasis, eczema, squamous cell carcinoma, acneiform eruptions caused by medications, steroid acne, steroid folliculitis, bacterial folliculitis, or any other facial disease or condition.
5. Excessive facial hair (i.e., heavy beard or mustache), facial tattoos, or facial disfigurement, excessive hair on the neck, upper chest, shoulders and upper back region that would interfere with study assessments.
6. Subjects with a serious and/or chronic medical condition such as chronic or active liver disease, renal impairment, heart disease, severe respiratory disease, rheumatoid arthritis, current malignancies, immunocompromised conditions, or any other disease that, in the opinion of the investigator, would interfere with the study or place the subject at unacceptable risk.
7. Subjects who have been treated for alcohol dependence or alcohol or drug abuse in the year prior to Baseline (Day 1).
8. Subjects who have been in another investigational trial within 30 days of Baseline (Day 1).
9. Subjects may not have a personal relationship with any member of the study staff or be part of the staff at the medical practice.
10. HIV Ag/Ab Combo, Hepatitis B (HBsAg (B)) and Hepatitis C (anti-HCV (C)) positive subjects.

Min Age: 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2017-10-04 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anirudh Gautam, Study Director — Dr. Reddy's Laboratories Inc.
Locations (2):
- United States (2):
  - Dr. DuBois, Austin, Texas
  - Dr. Jones, Austin, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- DFD-03 Lotion: DFD-03 Lotion was applied to the affected areas twice daily for 1 minute and rinsed off.
- Tazorac Cream: Tazorac Cream was applied to the affected areas once daily and left on for ~12 hours.
Period: Overall Study
Arm/Group | DFD-03 Lotion | Tazorac Cream
Started | 34 | 24
Completed | 32 | 21
Not Completed | 2 | 3
Not completed — Adverse Event | 0 | 2
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Population: The Intent to Treat (ITT) population comprised of all randomized subjects.
Groups:
- DFD-03 Lotion: DFD-03 Lotion were applied to the affected areas twice daily for 1 minute and rinsed off. Thirty four (34) subjects were enrolled into this arm, of whom 32 completed the study.
  Tazarotene Lotion, 0.1%: DFD-03 (Tazarotene Lotion, 0.1%) applied Twice Daily for 1 minute and rinsed off
- Tazorac Cream: Tazorac Cream were applied to the affected areas once daily and left on for ~12 hours. Twenty four (24) subjects were enrolled into this arm, of whom 21 completed the study.
  Tazarotene Cream, 0.1%: Tazorac® (tazarotene) Cream, 0.1% applied Once Daily and left for approximately 12 hours
- Total: Total of all reporting groups
Arm/Group | DFD-03 Lotion | Tazorac Cream | Total
Number analyzed (Participants) | 34 | 24 | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 17 (7) | 18 (5) | 18 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 12 | 28
  Male | 18 | 12 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 5 | 12
  Not Hispanic or Latino | 27 | 19 | 46
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 6 | 15
  White | 23 | 16 | 39
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 34 | 24 | 58
Body Mass Index (BMI) [Mean (Standard Deviation); unit: Kilograms per meter square] | 23.0 (4.4) | 28.1 (7.5) | 25.1 (6.4)

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Concentration (Cmax)
Description: The maximum plasma concentration of tazarotenic acid post dosing on Day 21 (Cmax(ss))
Time Frame: Day 21
Population: The Pharmacokinetic (PK) population included subjects who provided PK samples at all pre-specified time points.
Measure: Mean (Standard Deviation); unit: pg/mL
Groups:
- DFD-03 Lotion: DFD-03 Lotion was applied to the affected areas twice daily for 1 minute and rinsed off. Thirty four (34) subjects were enrolled into this arm, of whom 32 completed the study.
  Tazarotene Lotion, 0.1%: DFD-03 (Tazarotene Lotion, 0.1%) applied Twice Daily for 1 minute and rinsed off
- Tazorac Cream: Tazorac Cream was applied to the affected areas once daily and left on for ~12 hours. Twenty four (24) subjects were enrolled into this arm and 21 subjects completed the study.
  Tazarotene Cream, 0.1%: Tazorac® (tazarotene) Cream, 0.1% applied Once Daily and left for approximately 12 hours
Arm/Group | DFD-03 Lotion | Tazorac Cream
Number analyzed (Participants) | 32 | 21
pg/mL | 180.78 (50.0) | 529.91 (40.2)

2. Primary Outcome: Area Under the Curve (AUC0-24) at Steady State
Description: The Area Under the Curve time 0 to 24 hours (AUC0-24ss) of tazarotenic acid at steady state (Day 21)
Time Frame: Day 21
Population: The PK population included subjects who provided PK samples on Day 14 and Day 21.
Measure: Mean (Standard Deviation); unit: pg.hr/mL
Groups:
- Tazorac Cream: Tazorac Cream will be applied to the affected areas once daily and left on for ~12 hours. Twenty four (24) subjects were enrolled into this arm, of whom 21 completed the study.
  Tazarotene Cream, 0.1%: Tazorac® (tazarotene) Cream, 0.1% applied Once Daily and left for approximately 12 hours
Arm/Group | DFD-03 Lotion | Tazorac Cream
Number analyzed (Participants) | 32 | 21
pg.hr/mL | 4644.16 (43.6) | 8180.19 (38.6)

3. Primary Outcome: Number of Subjects With Treatment Emergent Adverse Events (TEAE)
Description: Number of subjects with at least one TEAE from the time of signing the consent until the end of the study (Approximately 21 days).
Time Frame: Day 1 to Day 21
Population: The Safety Population included all subjects randomized who provided at least one post baseline safety assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | DFD-03 Lotion | Tazorac Cream
Number analyzed (Participants) | 34 | 24
Participants | 34 | 23

4. Secondary Outcome: Time to Maximum Concentration (Tmax) of Tazarotenic Acid
Description: Time to maximum concentration (Tmax(ss)) of tazarotenic acid at steady state (Day 21)
Time Frame: Day 21
Population: The PK population included all subjects who provided PK samples at all pre-specified time-points.
Measure: Median (Full Range); unit: hours
Arm/Group | DFD-03 Lotion | Tazorac Cream
Number analyzed (Participants) | 32 | 21
hours | 4.02 [3.85 to 8.10] | 5.95 [4.00 to 8.10]

ADVERSE EVENTS:
Time Frame: From the time of study consent until end of treatment or treatment discontinuation (Approximately 21 days).
Description: Adverse event data were collected from the time the Informed Consent Form was signed until study product treatment was discontinued, except for spontaneously reported SAEs, which were to be reported up to 30 days after discontinuing study product use.
Arm/Group | DFD-03 Lotion | Tazorac Cream
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/24
Other Adverse Events (participants affected / at risk) | 34/34 | 23/24
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | DFD-03 Lotion (N=34) | Tazorac Cream (N=24)
Application site erythema (General disorders) | 33 | 21 — Erythema at the site of application
Application site exfoliation (General disorders) | 34 | 23 — Exfoliation of the skin at the application site
Application site dryness (General disorders) | 34 | 22 — Dryness of the skin at the site of application
Application site pain (General disorders) | 25 | 19 — Pain at the site of application
Application site pruritus (General disorders) | 25 | 17 — Pruritus at the site of application
Eczema Asteatotic (Skin and subcutaneous tissue disorders) | 5 | 0
Eczema (Skin and subcutaneous tissue disorders) | 2 | 1
Headache (Nervous system disorders) | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-02): https://cdn.clinicaltrials.gov/large-docs/93/NCT03599193/Prot_SAP_000.pdf